CLINICAL TRIAL: NCT02094430
Title: Clinical Pharmacology, Efficacy and Safety Study of FGTW in Paediatric Patients With Severe Congenital Fibrinogen Deficiency
Brief Title: Human Fibrinogen Concentrate (FGTW) in Pediatric Patients With Congenital Fibrinogen Deficiency
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGTW-1004
Record Dates: First submitted 2014-02-26; First posted 2014-03-21 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Hypofibrinogenemia, Congenital; Afibrinogenemia, Congenital
MeSH Terms: conditions — Afibrinogenemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FGTW (Experimental)
  Interventions: Drug: biological: human fibrinogen concentrate

INTERVENTIONS:
Drug: biological: human fibrinogen concentrate

SUMMARY:
The aim of the study is to evaluate clinical pharmacology, efficacy and safety of FGTW in pediatric patients with congenital fibrinogen deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form by parents or a legal representative
* Age less or equal to 12 years old
* Patients with inherited afibrinogenemia or severe inherited hypofibrinogenemia
* Negative results on HCG-based pregnancy test for females of childbearing potential (presence of menstruation)

Exclusion Criteria:

* Dysfibrinogenemia
* Acquired fibrinogen deficiency
* Suspected present or past anticoagulation inhibitor
* Personal history of venous or arterial thrombosis or thromboembolic event
* Co-morbidity with other/unrelated coagulopathies
* Administration of any fibrinogen concentrate or fibrinogen containing blood product during the last 15 days
* Permanent treatment with antithrombotic or anti-platelet agents such as heparins, anti-IIa or anti-Xa agents, aspirin, clopidogrel and NSAIDs.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Investigator's overall assessment of efficacy of FGTW on hemostasis using a 4-point scale at the end of each bleeding or surgical episode. | 6 hours or up to 5 days
Terminal half life for Fibrinogen antigen and activity | 5 days

SECONDARY OUTCOMES:
Adverse Events | Participants will be followed for the duration of their participation in the study, an expected average of 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- Hopital Necker enfants malades, Paris, France
- Hôpital Hôtel Dieu, Beirut, Lebanon
- Hôpital d'enfants - CHU Avicenne, Rabat, Morocco
- Faculty Ihsan Dogramaci Children's Hospital, Ankara, Turkey (Türkiye)